CLINICAL TRIAL: NCT04666415
Title: Monocentric Single-blind Randomized Controlled Trial Evaluating the Impact of the Addition of a Specific and Personalized Body Approach by Osteopathic Treatment in the Care of Adolescents With Anorexia Nervosa
Brief Title: Impact of the Addition of a Specific and Personalized Body Approach by Osteopathic Treatment in the Care of Adolescents With Anorexia Nervosa.
Acronym: ACAMTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY IMM-N°010-2019
Record Dates: First submitted 2020-08-28; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Anorexia Nervosa; Osteopathic Medicine
Keywords: Interoception; Randomized controlled trial; Body approach
MeSH Terms: conditions — Anorexia Nervosa | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor of the clinical and psychological outcomes (research psychologist) will be blinded to the treatment group and will use standardized research questionnaires. Assessors of the osteopathic outcomes will not perform the osteopathic sessions, to guarantee an independent evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic treatment + as-usual treatment (Experimental): Osteopathic treatment: a protocol of 5 sessions of osteopathic treatment that have a 25 minutes duration and are spaced of around one week between two sessions.
  As-usual treatment: The outpatient and inpatient treatment of the patients will be done in compliance with the Health Authorities' recommendations (HAS 2010). Multi-disciplinary care is proposed, possibly involving nurses, psychologists, psychiatrists, general practitioners, gynecologists, rheumatologists, dieticians, occupational therapists, body approach specialists and social workers.
  Interventions: Other: Osteopathic treatment
- As-usual treatment (No Intervention): As-usual treatment: The outpatient and inpatient treatment of the patients will be done in compliance with the Health Authorities' recommendations (HAS 2010). Multi-disciplinary care is proposed, possibly involving nurses, psychologists, psychiatrists, general practitioners, gynecologists, rheumatologists, dieticians, occupational therapists, body approach specialists and social workers.

INTERVENTIONS:
Other: Osteopathic treatment — Targeted osteopathic protocol for AN : 5 sessions of osteopathic treatment that are spaced around one week between 2 sessions. Soft specific palpatory techniques on the diaphragm, digestive system and cervical region will be realized during the session of 25 minutes.
  Arms: Osteopathic treatment + as-usual treatment

SUMMARY:
Abstract:

Background: Anorexia nervosa (AN) is a common pathology affecting mainly women (sex ratio 1/10), which starts most often during adolescence. The prognosis of the AN remains poor (10% of deaths and high risk of chronicity). Body dissatisfaction, disturbances in recognition and identification of body sensations are some of the key symptoms of AN. There is, however, a contrast between this consensual observation of the importance of troubles in body image in AN, and the relative deficit of specifically targeted body treatments. Our proposal for a body approach specifically dedicated to AN is based on the understanding that posture, breathing, muscle tension and body perception are closely linked to our psychological and emotional state, and are therefore disturbed in patients with AN.

The purpose of this monocentric randomized controlled trial is to evaluate if a targeted osteopathic protocol treatment for AN in addition to as-usual care is significantly more effective compared to as-usual care.

Methods: Seventy-two female patients meeting the inclusion criteria will be randomly assigned to one of the two treatment groups : one receiving the specific osteopathic treatment targeted for AN in addition to the as-usual care (group A) and the other one, the as-usual care (group B). The patients of group A will receive 5 sessions of osteopathic treatment for 25 minutes. Soft specific palpatory techniques on the diaphragm, digestive system and cervical region will be realized. The as-usual care is defined by the multidisciplinary approach recommended by the high authority of health. The primary outcome is the evaluation of interoceptive sensibility and secondary outcomes include clinical and psychopathology-related symptoms and assessment of somatic dysfonctions' evolution. A qualitative study will also be carried out, applying the Interpretative Phenomenological Analysis method. Patients will be included for a maximum of 14 weeks between the inclusion time and the last evaluation.

Discussion:

If the results of the study are positive (statistically significant effectiveness of this body approach in addition to as-usual care compared to as-usual treatment), patients with anorexia will be benefit from the possibility of additional treatment that is effective, relatively inexpensive, non-invasive and non-pharmacological.

ELIGIBILITY:
Inclusion Criteria:

* female
* patient aged between 13 to 20 years included
* patient has a Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-5) diagnosis of Nnorexia nervosa (restricting or binge-eating/purging types)
* Body Mass Index (BMI) ≥ 14 kg.m-²
* Followed up in consultation for at least 2 months or hospitalized in the psychiatry unit of Institut Mutualiste Montsouris
* has a clinical/somatic state compatible with the conduct of osteopathic treatment sessions (prior medical advice)
* is not in "separation period" (In the adolescent and young adult psychiatry department of Institut Mutualiste Montsouris, during a full-time hospitalization for AN, the "separation period" is linked to the establishment of a hospitalization contract between the medical team, the family and the patient. This contract will define a time of separation between the family and the patient. It is built around two axes: the final discharge weight allowing the patient to leave the service and the intermediate weight called "separation lifting weight". This lifting weight of separation is thus named because it puts an end to the first part of hospitalization that takes place in separation from the living environment of the patient (parents, friends, schooling...)
* signed the Informed Consent Form and both parents for minor patient,
* is not included in another research protocol.

Non-inclusion criteria:

* male
* patient under 13 years old or over 20 years old
* has contraindication to osteopathic body approach sessions (fracture, recent surgery, etc.)
* with a Body Mass Index (BMI) < 14 kg.m-²
* patient needs a naso-gastric tube
* is in "separation period"
* is not fluent in French
* is not covered by health insurance
* is included in another research protocol.

Exclusion criteria:

* patient has contraindication to osteopathic body approach sessions (fracture, recent surgery, somatic state not compatible with the osteopathic treatment)
* is not covered by health insurance
* is included in another research protocol.

Ages: 13 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the evolution of interoceptive sensitivity | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  fMAIA scale : Multidimensional Assessment of Interoceptive Awareness, French version
To evaluate the evolution of interoceptive sensitivity | Arm 1: Before the 3rd session of osteopathic treatment, Arm 2: 3 weeks after the first questionnaires
  fMAIA scale : Multidimensional Assessment of Interoceptive Awareness, French version
To evaluate the evolution of interoceptive sensitivity | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  fMAIA scale : Multidimensional Assessment of Interoceptive Awareness, French version

SECONDARY OUTCOMES:
To evaluate the evolution of weight | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  Weight measured in kilograms
To evaluate the evolution of weight | Arm 1: Before the 3rd session of osteopathic treatment, Arm 2: 3 weeks after the first questionnaires
  Weight measured in kilograms
To evaluate the evolution of weight | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  Weight measured in kilograms
To evaluate the presence of any physical pain | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  Actual physical pain (yes/no), precision of the localisation and intensity by Visual Analog Score (from 0 to 10)
To evaluate the presence of any physical pain | Arm 1: Before the 3rd session of osteopathic treatment, Arm 2: 3 weeks after the first questionnaires
  Actual physical pain (yes/no), precision of the localisation and intensity by Visual Analog Score (from 0 to 10)
To evaluate the presence of any physical pain | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  Actual physical pain (yes/no), precision of the localisation and intensity by Visual Analog Score (from 0 to 10)
To evaluate the presence of constipation | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  Any constipation (yes/no) and precision of number of bowel movements per week
To evaluate the presence of constipation | Arm 1: Before the 3rd session of osteopathic treatment, Arm 2: 3 weeks after the first questionnaires
  Any constipation (yes/no) and precision of number of bowel movements per week
To evaluate the presence of constipation | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  Any constipation (yes/no) and precision of number of bowel movements per week
To evaluate the evolution of nature of patient's eating disorder symptoms | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  EDDS : Eating Disorder Diagnostic Scale. Self-reported questionnaire for diagnosis of eating disorders.
To evaluate the evolution of nature of patient's eating disorder symptoms | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  EDDS : Eating Disorder Diagnostic Scale. Self-reported questionnaire for diagnosis of eating disorders.
To evaluate the evolution of seriousness of patient's eating disorder symptoms | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  EDI-2: Eating Disorders Inventory. The EDI-2 total score ranges from 91 to 546. Higher score means a worse outcome.
To evaluate the evolution of seriousness of patient's eating disorder symptoms | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  EDI-2: Eating Disorders Inventory. The EDI-2 total score ranges from 91 to 546. Higher score means a worse outcome.
To evaluate the evolution of seriousness of concerns about body image | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  BSQ: Body shape questionnaire. The BSQ score ranges from 34 to 204. Higher score means a worse outcome.
To evaluate the evolution of seriousness of concerns about body image | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  BSQ: Body shape questionnaire. The BSQ score ranges from 34 to 204. Higher score means a worse outcome.
To evaluate the evolution of seriousness of alexithymia | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  BVAQ-B: Bermond-Vorst Alexithymia Questionnaire Form B. The BVAQ-B score ranges from 20 to 100. Higher score means a worse outcome.
To evaluate the evolution of seriousness of alexithymia | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  BVAQ-B: Bermond-Vorst Alexithymia Questionnaire Form B. The BVAQ-B score ranges from 20 to 100. Higher score means a worse outcome.
To evaluate the evolution of seriousness of self-esteem | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  RSE: Rosenberg Self-esteem Scale. The RSE score ranges from 10 to 40. Higher score means a worse outcome.
To evaluate the evolution of seriousness of self-esteem | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  RSE: Rosenberg Self-esteem Scale. The RSE score ranges from 10 to 40. Higher score means a worse outcome.
To evaluate the evolution of seriousness of anxiety | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  STAI-Y: State-Trait Anxiety Inventory, Form Y. The STAI-Y score ranges from 20 to 80. Higher score mean a worse outcome.
To evaluate the evolution of seriousness of anxiety | Arm 1: Before the 3rd session of osteopathic treatment, Arm 2: 3 weeks after the first questionnaires
  STAI-Y: State-Trait Anxiety Inventory, Form Y. The STAI-Y score ranges from 20 to 80. Higher score mean a worse outcome.
To evaluate the evolution of seriousness of anxiety | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  STAI-Y: State-Trait Anxiety Inventory, Form Y. The STAI-Y score ranges from 20 to 80. Higher score means a worse outcome.
To evaluate the evolution of seriousness of depressive experiences | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  DEQ: Depressive Experiences Questionnaire - Adolescent Version. The Depressive Experiences Questionnaire (DEQ) is a 66 item questionnaire where participants rate themselves on life experiences and personality characteristics frequently associated with depression. Participants are asked to rate each item on a seven-point Likert-type scale ranging from strongly disagree (1) to strongly agree (7). Analysis of results produces 3 factors: Dependency, Self-criticism, and Efficacy.
To evaluate the evolution of seriousness of depressive experiences | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  DEQ: Depressive Experiences Questionnaire - Adolescent Version. The Depressive Experiences Questionnaire (DEQ) is a 66 item questionnaire where participants rate themselves on life experiences and personality characteristics frequently associated with depression. Participants are asked to rate each item on a seven-point Likert-type scale ranging from strongly disagree (1) to strongly agree (7). Analysis of results produces 3 factors: Dependency, Self-criticism, and Efficacy.
To evaluate the evolution of seriousness of depression | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  HAD-depression: Hospital Anxiety and Depression scale-depression. The HAD-depession score ranges from 0 to 21. Higher score means a worse outcome.
To evaluate the evolution of seriousness of depression | Arm 1: Before the 3rd session, Arm 2: 3 weeks after the first questionnaires
  HAD-depression: Hospital Anxiety and Depression scale-depression. The HAD-depession score ranges from 0 to 21. Higher score means a worse outcome.
To evaluate the evolution of seriousness of depression | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  HAD-depression: Hospital Anxiety and Depression scale-depression. The HAD-depession score ranges from 0 to 21. Higher score means a worse outcome.
To evaluate the evolution of nature and seriousness of self-injury | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  OSI: Ottawa Self-injury Questionnaire. OSI (Ottawa Self-Injury) to measure occurrence, frequency, level of motivation to stop, types and functions and potential addictive features of self-injury
To evaluate the evolution of nature and seriousness of self-injury | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  OSI: Ottawa Self-injury Questionnaire. OSI (Ottawa Self-Injury) to measure occurrence, frequency, level of motivation to stop, types and functions and potential addictive features of self-injury
To evaluate the evolution of quality of life | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  ED-QOL: Eating Disorders Quality of Life Scale. The EDQOL has 25 items that contribute to four subscales (Psychological, Physical/Cognitive, Work/School, and Financial), which combined produce an overall quality of life score. Each item is coded on a five-point scale and asks the participant to rate the extent to which they perceive their eating disorder to affect their quality of life in different domains. Higher scores indicate lower quality of life.
To evaluate the evolution of quality of life | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  ED-QOL: Eating Disorders Quality of Life Scale. The EDQOL has 25 items that contribute to four subscales (Psychological, Physical/Cognitive, Work/School, and Financial), which combined produce an overall quality of life score. Each item is coded on a five-point scale and asks the participant to rate the extent to which they perceive their eating disorder to affect their quality of life in different domains. Higher scores indicate lower quality of life.
To evaluate the evolution of seriousness of physical activity dependence | Arm 1: 3 weeks after inclusion ie 1 week before the first session, Arm 2: 3 weeks after inclusion
  EDS-R: Exercise-Dependence Scale-Revised, The EDS-R score ranges from 21 to 126. Higher score means worse outcome
To evaluate the evolution of seriousness of physical activity dependence | Arm 1: Before the 3rd session, Arm 2: 3 weeks after the first questionnaires
  EDS-R: Exercise-Dependence Scale-Revised, The EDS-R score ranges from 21 to 126. Higher score means worse outcome
To evaluate the evolution of seriousness of physical activity dependence | Arm 1: 1 week after the 5th session of osteopathic treatment, Arm 2: 6 weeks after the first questionnaires
  EDS-R: Exercise-Dependence Scale-Revised, The EDS-R score ranges from 21 to 126. Higher score means worse outcome
To evaluate the evolution of somatic dysfonctions (for Arm 1) | Arm 1: before each of the 5 osteopathic treatment sessions
  SOAP note form. This is a standardized tool to evaluate somatic dysfunctions (sensitivity, mobility, texture, asymmetry) and severity (from 0 to 3) for each body region
To evaluate the evolution of somatic dysfonctions (for Arm 1) | Arm 1:1 week after the 5th session of osteopathic treatment
  SOAP note form. This is a standardized tool to evaluate somatic dysfunctions (sensitivity, mobility, texture, asymmetry) and severity (from 0 to 3) for each body region

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie LETRANCHANT, M.D., Principal Investigator — Institut Mutualiste Montsouris; Maurice CORCOS, M.D., Ph.D., Study Director — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Letranchant A, Montebello YK, Bigre CD, Wagner A, Curt F, Silva J, Nicolas I, Votadoro P, Kalindjian N, Korchonnoff A, Gutierre A, Novelli AB, Pham-Scottez A, Corcos M. The ACAMTO study-impact of add-on osteopathic treatment on adolescent patients with anorexia nervosa: study protocol for a randomized controlled trial. Trials. 2021 Nov 24;22(1):839. doi: 10.1186/s13063-021-05810-8. PMID 34819116